CLINICAL TRIAL: NCT02094950
Title: Acupuncture Feasibility Trial for Dyspnea in Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: UPCC 11513
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer; Dyspnea
Keywords: concurrent chemotherapy; concurrent radiation
MeSH Terms: conditions — Lung Neoplasms; Dyspnea | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lung Cancer Patient with Dyspnea (Experimental)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
This is a single arm clinical trial to establish the feasibility of conducting a clinical trial of acupuncture in reducing dyspnea among lung cancer survivors who have completed chemoradiotherapy. Twelve subjects with dyspnea will be recruited to this clinical trial. Up to 10 sessions of acupuncture will be delivered over the course of 8-10 weeks. The primary outcome will be dyspnea as measured by the English version of the Cancer Dyspnea Scale at the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lung Cancer (Non small cell and small cell both eligible)
* Completion of concurrent CRT at least 6 months prior to randomization.
* Dyspnea which worsened after Chemoradiotherapy, leading to a ATS dyspnea score greater than or equal to 2 (Walks slower than people of the same age on the level because of breathlessness or has to stop for breath when walking at own pace on level)
* Ability to understand written English -Willingness to adhere to all study-related procedures
* Age 18 years old
* ECOG Performance Status 1-3

Exclusion Criteria:

* Current receipt of therapy for treatment related pneumonitis for 3 weeks.
* Surgical resection of this LC (lobectomy or pneumonectomy)
* Another organic cause of dyspnea necessitating treatment (eg pleural effusion appropriate for thoracentesis, rapidly progressive intrathoracic recurrence, symptomatic pulmonary embolus after CRT, untreated anemia with hemoglobin8 g/dL)
* Current bleeding disorder by history
* Life expectancy of 12 weeks, as assessed by primary oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bauml, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States